CLINICAL TRIAL: NCT01905904
Title: The Comparision of Different Doses of Sevoflurane for Induction of General Anesthesia in Electroconvulsive Therapy
Brief Title: Sevoflurane in Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, assistant profesor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ulkü_2
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: ECT; Anesthesia
Keywords: electroconvulsive therapy; seizures; sevoflurane
MeSH Terms: conditions — Seizures | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevorane (Active Comparator): Sevorane 4% concentration during anesthesia induction
  Interventions: Drug: sevorane
- sevorane %7 (Active Comparator): Sevorane 7% concentration during anesthesia induction
  Interventions: Drug: sevorane

INTERVENTIONS:
Drug: sevorane — Sevorane 4% Sevorane 7%
  Other Names: Sevoflurane

SUMMARY:
The purpose of the study was to investigate the effects of different doses of sevoflurane used in electroconvulsive therapy (ECT) on duration of seizure, hemodynamic response and recovery profiles

DETAILED DESCRIPTION:
Motor (EMG) and electroencephalography seizure duration (EEG), heart rate (HR) and mean arterial pressure (MAP) values, and recovery times were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Study included 25 patients of American Society of Anesthesiologists (ASA) physical status I-II aged between 18-60 years who were scheduled for ECT sessions under general anesthesia

Exclusion Criteria:

* Pregnancy
* Cerebrovascular disease
* Epilepsy
* Unstable cardiovascular disease
* Chronic obstructive pulmonary disease; and
* Renal or hepatic failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
sevoflurane used in electroconvulsive therapy (ECT) on duration of seizure | taken prior to the seizure

SECONDARY OUTCOMES:
sevoflurane used in electroconvulsive therapy (ECT) on hemodynamic response. | taken prior to the seizure

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Toprak, Professor, Principal Investigator — Inonu University
Locations (1):
- Inonu Unıversity School of Medicine, Malatya, Turkey (Türkiye)